CLINICAL TRIAL: NCT06997042
Title: Creation of Arteriovenous Fistulas for Hemodialysis Using the End-to-side Anastomotic Technique vs. Piggyback. Randomized Clinical Trial
Brief Title: Creation of Arteriovenous Fistulas for Hemodialysis Using the End-to-side Anastomotic Technique vs. Piggyback.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Adrián López, Medical Doctor, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCB/2025/0087
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis
Keywords: hemodialysis; vascular access; arteriovenous fistula; piggyback
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terminolateral anastomosis (Placebo Comparator): Patients assigned to this arm of intervention will have an anastomosis performed with the terminolateral anastomosis technique described in the protocol.
  Interventions: Procedure: Terminolateral anastomotic technique
- Piggyback anastomosis (Active Comparator): Patients assigned to this arm of intervention will be have an anastomosis performed with the piggyback anastomosis technique described in the protocol.
  Interventions: Procedure: Piggyback anastomotic technique

INTERVENTIONS:
Procedure: Terminolateral anastomotic technique — Suturing the vein and artery of the arteriovenous fistula with a terminolateral anastomotic suture.
  Arms: Terminolateral anastomosis
Procedure: Piggyback anastomotic technique — Suturing the vein and artery of the arteriovenous fistula with a piggyback anastomotic technique.
  Arms: Piggyback anastomosis

SUMMARY:
This study is designed to compare two surgical techniques used to create arteriovenous fistulas (AVFs), which are necessary for hemodialysis in patients with advanced chronic kidney disease (CKD). AVFs are preferred over other forms of vascular access because they last longer and have fewer complications. However, many AVFs fail to mature properly, making them unusable for dialysis.

The two techniques being studied are the traditional End-to-Side (ETS) method and a newer technique called Piggyback Straight Line Onlay Technique (pSLOT). Early studies suggest that pSLOT may reduce complications like narrowing (stenosis), clotting (thrombosis), and failure of the AVF, but more robust data from randomized clinical trials is needed.

Patients aged 18 or older with stage 4 or 5 CKD, who are eligible for a new AVF and meet health criteria, may participate. During the operation, participants are randomly assigned to receive either the ETS or pSLOT technique. The procedure is done under local or regional anesthesia. Follow-up appointments are scheduled at 1 and 12 months to assess fistula maturation, blood flow, and whether it can be successfully used for dialysis. Remote follow-ups are allowed if needed.

Participation is voluntary, requires informed consent, and all data is kept strictly confidential. The study follows national and international ethical standards and has been approved by an ethics committee.

DETAILED DESCRIPTION:
Creation of Arteriovenous Fistulas for Hemodialysis: End-to-Side vs. Piggyback Anastomosis - A Randomized Clinical Trial

1. Background and Rationale

   Chronic Kidney Disease (CKD) affects an estimated 15.1% of the Spanish population and is a growing public health concern, especially due to its progression to advanced stages requiring renal replacement therapy (RRT). Hemodialysis is the most common RRT, and the quality of vascular access significantly influences outcomes in these patients.

   Among vascular access options, arteriovenous fistulas (AVFs) are preferred over central venous catheters (CVCs) and arteriovenous grafts (AVGs), due to superior durability, fewer complications, and lower hospitalization rates. However, AVFs suffer from high early failure rates, with maturation failures occurring in up to 60% of cases.

   Traditionally, the end-to-side (ETS) anastomosis is the gold standard for AVF creation. In recent years, an alternative technique called the Piggyback Straight Line Onlay Technique (pSLOT) has shown potential benefits, including improved hemodynamics, reduced stenosis, and lower rates of thrombosis and dysfunction.

   Despite promising retrospective data and small prospective studies, no robust randomized controlled trial has conclusively determined whether pSLOT offers superior outcomes compared to the classical ETS technique.
2. Study Hypothesis

   The null hypothesis is that there will be no significant difference between ETS and pSLOT techniques in terms of:
   * Clinical and ultrasound-based maturation at 1 month
   * Clinical and ultrasound-based maturation, patency, and functionality at 12 months
3. Study Objectives

   Primary Objective

   To compare the rate of clinical and ultrasonographic maturation at 1 month, and the combined rate of maturation, patency, and functionality at 12 months between ETS and pSLOT groups.

   Secondary Objectives

   To compare:
   * Juxta-anastomotic stenosis rate
   * Thrombosis rate
   * Reintervention rate
   * Fistula blood flow
   * Maturation and surgery times
   * Wound-related complications
4. Methods and Study Design

   This is a single-center, prospective, randomized, controlled trial with two parallel groups:
   * Group A: ETS technique
   * Group B: pSLOT technique

   Randomization occurs intraoperatively (1:1 allocation) using a centralized system. The patient is blinded to the allocation. The surgical team is not blinded due to the nature of the procedure, and follow-up staff are aware of the technique due to its visibility on ultrasound.

   The trial will enroll 130 patients to account for a 15% dropout rate, aiming for 56 evaluable patients per group. This sample size is based on previous data indicating differences in juxta-anastomotic stenosis rates (16.7% vs. 40.3%).
5. Inclusion and Exclusion Criteria

   Inclusion
   * Adults ≥18 years
   * CKD stage 4 or 5 (pre-dialysis or on hemodialysis)
   * Anatomically suitable for native AVF creation
   * No prior AVFs in the same or proximal site
   * Informed consent provided

   Exclusion
   * Pregnant women
   * Life expectancy <1 year
   * Central vein stenosis or occlusion
   * Known coagulopathy, active infection, or severe systemic disease
   * Scheduled kidney transplant within 60 days
   * Previous upper extremity vascular surgery in the planned site
6. Procedure and Follow-Up

   Preoperative Assessment
   * Clinical history and physical examination
   * Duplex ultrasound mapping of arteries and veins in both upper limbs
   * Eligibility based on standard anatomical criteria
   * Consent obtained post-screening

   Surgical Procedure
   * Performed under local/regional anesthesia
   * Intraoperative data: type of fistula (distal/proximal), duration, success, Doppler flow, diameter, and complications

   Follow-up Visits
   * 1 Month: Clinical and Doppler ultrasound to assess maturation and flow
   * 12 Months: Same assessments plus record of any interventions or complications

   Remote follow-up may be permitted if patients cannot attend physically.
7. Definitions of Key Outcomes

   * Clinical Maturation: Fistula suitable for two-needle cannulation and achieving dialysis flow
   * Ultrasound Maturation: Diameter >5mm, depth <5mm, and flow >500 ml/min
   * Functionality: Used for regular dialysis with adequate flow
   * Patency: Defined as primary, assisted primary, or secondary per European Vascular Society guidelines
8. Statistical Analysis

   * Software: SPSS v23
   * Descriptive statistics for demographics and clinical variables
   * Chi-square for proportions
   * Kaplan-Meier survival curves and log-rank test for time-to-event analysis
   * Multivariate regression for confounders: age, sex, diabetes, vessel diameter, fistula location

   Significance threshold: p < 0.05
9. Ethics and Regulatory Aspects

   * Protocol complies with Declaration of Helsinki (2013) and Spanish Biomedical Research Law (14/2007)
   * Approved by institutional ethics committee
   * Data anonymized and managed per EU Regulation 2016/679
   * Participation is voluntary, with informed consent required

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Able to meet protocol requirements, including follow-up.
* Incident or prevalent patient with advanced chronic kidney disease in the hemodialysis stage (stage 5D).
* In predialysis patients (stage 5), if renal replacement therapy (hemodialysis) is anticipated to be required within the next 6 months (based on standard clinical criteria).
* Who, based on their associated pathology and according to medical criteria, can withstand the initial surgery and arteriovenous access maintenance procedures.
* Have a current ultrasound with preoperative venous and arterial mapping.
* Meet the anatomical requirements for AVF creation:

  * Wrist: artery >2 mm, vein >2 mm in diameter
  * Elbow: artery >3 mm, vein >3 mm in diameter
  * Absence of arterial calcification or occlusion, or other aberrant arterial anatomy.
  * Adequate arterial and venous patency.
  * Vein-to-skin distance <5 mm.
* Candidate for creation of a native arteriovenous fistula for hemodialysis, either distal (radiocephalic) or proximal (humerocephalic or humerobasilic).
* No immediate transplant scheduled within the next 60 days (inclusion on the kidney transplant waiting list is not a contraindication for entry into the study, nor for the creation of an arteriovenous fistula).
* No prior arteriovenous surgeries in the same or proximal location.
* Correct understanding of the study conditions and acceptance to participate.

Exclusion Criteria:

* Pregnant women.
* Life expectancy <1 year.
* Arteriovenous prostheses (non-native fistulas), previous arteriovenous fistula repairs, arteriovenous accesses created in the lower extremities, and unusual (exotic) accesses.
* Known or suspected central venous stenosis/occlusion on the side of the planned access.
* Repair of previous arteriovenous accesses (proximal reanastomoses).
* Biological immunosuppression.
* History or evidence of serious systemic illness, including:

  * Cardiac disease (New York Heart Association functional class III or IV, as evidenced by the inability to lie still), myocardial infarction within 6 weeks prior to randomization, ventricular tachyarrhythmia requiring ongoing treatment, or unstable angina.

Suspected or documented hypercoagulable or hypocoagulable state or Clinically significant active infection (White blood count > 15,000 cells/mm3) other than the use of a treated CVC.

* Any other condition that, in the investigator's judgment, prevents an adequate evaluation of the safety and efficacy of the study or poor compliance.
* Patient unwilling or unable to attend follow-up follow-ups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of clinical and echographic maduration of the fistula | 1 month and 12 months

SECONDARY OUTCOMES:
Percentage juxta-anastomotic stenosis, thrombosis, reinterventions, fistula flow, maduration time, surgical time, wound complications | 1 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaspar Mestres, Medicine, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share individual participant data (IPD) from this study with other qualified researchers. Shared data will include anonymized information related to demographics, surgical technique, AVF maturation, complications, and follow-up outcomes. Data will be available upon reasonable request after publication and with approval from the study investigators, in compliance with ethical guidelines and data protection regulations.
Supporting Information: Study Protocol
Time Frame: 1 year after publication, during 5 years.
Access Criteria: Upon reasonable request, qualified researchers will be able to access to anonymized data of the study.